CLINICAL TRIAL: NCT05898971
Title: Effect of Robotic Hand Versus Mirror Therapy on Hand Functions in Stroke Patients
Brief Title: Robotic Hand on Hand Functions in Strokes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Batterjee Medical College (Other)
Responsible Party: Principal Investigator, Mariam Elsayed Mohamed Abd Alaal, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BMC
Record Dates: First submitted 2023-05-21; First posted 2023-06-12 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2023-09

CONDITIONS: CVA (Cerebrovascular Accident)
Keywords: Stroke; Hand Grip Strength
MeSH Terms: conditions — Stroke | interventions — Robotics

STUDY DESIGN:
Intervention Model Description: Randomized Comparative trial
Who Masked: Outcomes Assessor
Masking Description: single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): received robotic gloves training
  Interventions: Other: Robotic
- Group B (Experimental): received mirror therapy
  Interventions: Other: Mirror

INTERVENTIONS:
Other: Robotic — Patients receive robotic training (grasp and grip)
  Arms: Group A
Other: Mirror — Patients receive mirror therapy
  Arms: Group B

SUMMARY:
robotic glove training could be a useful aid for these patients. The aim of this study was to investigate the effect of Robotic gloves versus mirror therapy on Hand function in patients with cerebral vascular accident .

DETAILED DESCRIPTION:
Post stroke patients aged over 40 years were randomly assigned into three groups (A and B ) Group . Maximum hand grip strength, Hand and Fugl-Meyer Assessment-Upper Extremity (FMA-UE), were assessed at baseline, post-intervention, and six-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

Spasticity level 1 or 1+ according to modified Ashworth scale

Exclusion Criteria:

Uncontrolled seizures hand fractures or surgery

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
hand grip strength | 8 weeks, and six-month follow-up.
  Hand Dynamometer will be used to evaluate the hand's grip strength
Hand manual function | 8 weeks, and six-month follow-up.
  Box and block test for measuring the manual dexterity of patients

SECONDARY OUTCOMES:
Fugl-Meyer Assessment-Upper Extremity (FMA-UE) | 8 weeks, and six-month follow-up.
  It evaluates sensorimotor impairment

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Mariam Salem, Principal Investigator — Professor of Physical Therapy , Batterjee Medical College.
Locations (1):
- Dr. Mariam Salem, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No